CLINICAL TRIAL: NCT02120235
Title: Investigating Lysosomal Storage Diseases in Minority Groups
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: O & O Alpan LLC (Other)
Responsible Party: Sponsor
Other Study IDs: 14-CFCT-11
Record Dates: First submitted 2014-04-17; First posted 2014-04-22 (Estimated); Last update posted 2017-04-04 (Actual); Status verified 2017-04

CONDITIONS: Lysosomal Storage Disorders; Gaucher Disease; Fabry Disease; Pompe Disease; Niemann-Pick Disease
Keywords: Lysosomal storage disorders; LSD; Gaucher disease; Fabry disease; Pompe disease; Niemann-Pick disease
MeSH Terms: conditions — Lysosomal Storage Diseases; Gaucher Disease; Fabry Disease; Glycogen Storage Disease Type II; Niemann-Pick Diseases

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Biospecimen Retention: Samples With DNA — Blood

SUMMARY:
Although lysosomal storage disorders, such as Fabry disease, Gaucher disease, and Pompe disease, represent serious challenges in the healthcare system, no study has yet investigated the prevalence of these diseases in the US. Frequently, patients show progressive worsening of symptoms for several years before they get diagnosed. Since many of these diseases can be managed therapeutically, it is important to identify and treat patients in order to avoid organ damage. The investigators aim to undertake a screening study that identifies undiagnosed patients with lysosomal storage disorders and determine the prevalence of these diseases with special focus on underrepresented minority groups.

ELIGIBILITY:
Inclusion Criteria:

* Subject is greater than or equal to 1 day of age and less than or equal to 100 years of age
* Subject is managed by a physician in the Washington, D.C metro area
* Subject is getting blood work as part of standard clinical care and there is at least 60 uL blood remained in a tube after all clinical tests were run

Exclusion Criteria:

* Absolute contraindication for blood drawing
* Subject cannot be traced back by the referring physician upon a positive screening result

Ages: 1 Day to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The study population will comprise of patients of healthcare institutions in the Washington, D.C. metro area .
Sampling Method: Non-Probability Sample
Enrollment: 20000 (Estimated)
Dates: Start 2014-02; Primary Completion 2018-02 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Number of patients identified with lysosomal storage disorders | 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- O&O Alpan, LLC, Fairfax, Virginia, United States